CLINICAL TRIAL: NCT06172517
Title: Impact of Plantar Orthosis on Postural Control and Gait in Individuals With Plantar Fasciopathy
Brief Title: Plantar Fasciitis Management on Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Responsible Party: Principal Investigator, Rubens da Silva, Director and professor, Université du Québec à Chicoutimi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-404
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Rehabilitation; Aging Problems; Foot Diseases; Mobility Limitation
Keywords: Postural control; plantar orthoses; plantar fasciopathy; Biomechanics; Gait; Pain
MeSH Terms: conditions — Foot Diseases; Mobility Limitation; Pain

STUDY DESIGN:
Intervention Model Description: Clinical intervention by orthoses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Othesis intervention (Experimental): This group with custom-made foot orthotics prescribed by podiatrists (foot impression, polypropylene orthotics and covering at podiatrists' discretion).
  Interventions: Other: Orthosis intervention
- Control group (No Intervention): Without orthesis prescriptions by podiatrists.

INTERVENTIONS:
Other: Orthosis intervention — Clinical feasibility trial with one group using a custom-made foot orthotics prescribed by podiatrists (foot impression, polypropylene orthotics and covering at podiatrists' discretion).
  Arms: Othesis intervention

SUMMARY:
Foot pain is common in the general population. Plantar fasciopathy may affect 7% of the population at some time in their lives, but the incidence increases with age. This plantar problem is characterized by severe pain under the foot (at plantar level), which can be very incapacitating and disabling. This can lead to absenteeism from work, particularly for employees working in a standing posture. Various therapeutic avenues can be used to reduce pain and improve functionality, such as physiotherapy, infiltrations and surgery. In this research project, the propose the use of a conservative approach through the use of foot orthoses, which appears to be effective in reducing pain. The aim of the study is thus to better understand the effect of foot orthoses on postural balance and walking in workers with plantar fasciopathy. Participants will be assessed at baseline and eight weeks later to observe measured changes and clinical improvements following orthotic wear. Balance and gait pattern will be assessed using technological tools that have been validated in this respect. Participants will also be asked about their pain intensity. The hypothesis is that wearing the orthosis will improve the participants' balance and walking abilities, as well as reduce the level or intensity of their pain. In addition, this study could have an impact on the rate of absenteeism from work from current context of labour shortages.

DETAILED DESCRIPTION:
Plantar fasciopathy is a musculoskeletal disorder, known as a degeneration of the plantar fascia associated with a sensation of pain at plantar level. This disorder, for which around 2 million people a year receive treatment, has a prevalence of 3.6% to 7%, affecting both men and women between the ages of 45 and 64, and increasing with age. People aged between 25 and 65, who make up the majority of the working population, present 83% of plantar fasciopathy cases. According to CNESST statistics for 2022, 15,310 files opened concerned musculoskeletal disorders of the lower limb, 2133 of which involved the feet. There is also evidence of a possible cause-effect relationship between the number of hours spent standing or walking and the risk of developing plantar fasciopathy, which is indeed a major risk factor for many active workers. People with plantar fasciopathy will be absent from work more regularly, contributing to lower productivity at work. In addition to reduced work productivity, the cost of treatment has been estimated at US$584 million in the United States alone. In addition to pain, other deficits can be observed in people with plantar fasciopathy. A recent study also demonstrated its impact from a biomechanical point of view, notably on postural balance and gait in young adults suffering from this health problem. A number of treatments are currently used to treat this clinical foot condition, both conservatively and surgically. Among the most widely used conservative treatments, foot orthoses have been shown to be effective in reducing pain, despite the paucity of studies on the issue. Some studies have also demonstrated its effects on balance measures. Or, balance afferents originate from the somatosensory system, and tendon vibration can disrupt this system. However, few studies have measured its effects on postural control reactions via tendon vibration following orthotic use and in an ageing population, and no study has specifically investigated the effect of plantar orthoses in cases of plantar fasciopathy on gait pattern parameters in ageing workers.

ELIGIBILITY:
Inclusion Criteria:

* Present a history of pain under the heels for more than 3 months
* Have a diagnosis of plantar fasciopathy
* Pain of at least 3/10 under the heel
* Have post-static dyskinesia
* To be in the job market (adults between 20 and 65 years)

Exclusion Criteria:

* Severe systemic diseases
* Red flags (e.g. tumors),
* Musculoskeletal deformities affecting the lower limbs
* Musculoskeletal surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Postural control measures | baseline,immediate only for experimental group), and after 8 weeks.
  The participants will perform two 30-second trials on a strength platform (model BIOMEC400), the following tasks: without muscular vibration, with bilateral Achilles tendon vibration (Techno® concept VibrasensTM, France) in bipodal posture, and a balance task in semi-tandem posture with eyes open and closed. The vibration frequency chosen for the regions (sural triceps) will be 80 Hz. Center of Pressure (CoP) metrics will be used as main outcome such as sway CoP velocity variable (cm/s).
Gait measures | baseline,immediate only for experimental group), and after 8 weeks.
  The participants will be asked to walk at normal, slow and fast speeds on a GaitRite treadmill (GAI-TRite® Platinum Plus System 16' - 4.876 m, SN: Q209, CIR Systems Inc., Franklin, NJ, USA). Participants will perform each task twice.Main gait parameters will be used as main outcomes such as velocity in m/s.

SECONDARY OUTCOMES:
Ankle mobility and foot position measure | baseline and after 8 weeks.
  Ankle mobility will be measured using the Weight-Bearing Lunge Test will be used to assess foot positioning.
Lower Extremity Functional measure | baseline and after 8 weeks.
  The Lower Extremity Functional Scale(LEFS) questionnaire will be used to measure participants' level of functionality in the lower limbs. The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention. The columns on the scale are summed to get a total score. The maximum score is 80. he lower the score the greater the disability. The minimal detectable change is 9 scale points.
Pain measure by Foot function index | baseline and after 8 weeks.
  Foot Function Index will be used to measure foot pain and functionality. This index consists of 23 self-reported items divided into 3 subcategories: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
  The activity limitation subcategory consists of 5 items and measures limitations in activities because of foot problems, such as staying in bed all day. Recorded on a visual analogue scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain. Both total and subcategory scores are calculated.
Pain duration | baseline and after 8 weeks.
  In addition to sef-reported pain intensity and duration in number of months will calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens da Silva, PhD, Study Director — Université du Québec à Chicoutimi
Locations (1):
- Rubens da Silva, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan JR, Potter CB, Cappellini MD, Kurtz JB, Anderson MJ, Weatherall DJ. Aplastic crisis due to parvovirus infection in pyruvate kinase deficiency. Lancet. 1983 Jul 2;2(8340):14-6. doi: 10.1016/s0140-6736(83)90005-3. PMID 6134886
- [Background] Beeson P. Plantar fasciopathy: revisiting the risk factors. Foot Ankle Surg. 2014 Sep;20(3):160-5. doi: 10.1016/j.fas.2014.03.003. Epub 2014 Mar 22. PMID 25103701
- [Background] Ichioka T, Tashiro T, Hara T, Ichioka E. [Trial testing of the auto-refractometer NIDEK AR-3000 for mass examination of children and kindergarten, primary, junior high, and high school students]. Josai Shika Daigaku Kiyo. 1985;14(1):139-47. No abstract available. Japanese. PMID 3866618
- [Background] Richer L, Fortin E, Gagnon G, Ngomo S, Fernandes KBP, Cortis C, Sobczak S, da Silva RA. Impact of plantar fasciitis on postural control and walking in young middle-aged adults. Foot (Edinb). 2022 Dec;53:101951. doi: 10.1016/j.foot.2022.101951. Epub 2022 Nov 4. PMID 36463613
- [Background] Crawford F, Thomson CE. WITHDRAWN. Interventions for treating plantar heel pain. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000416. doi: 10.1002/14651858.CD000416.pub2. PMID 20091508
- [Background] Goguel V, Rosbash M. Splice site choice and splicing efficiency are positively influenced by pre-mRNA intramolecular base pairing in yeast. Cell. 1993 Mar 26;72(6):893-901. doi: 10.1016/0092-8674(93)90578-e. PMID 8458083
- [Background] Anderson J, Stanek J. Effect of foot orthoses as treatment for plantar fasciitis or heel pain. J Sport Rehabil. 2013 May;22(2):130-6. doi: 10.1123/jsr.22.2.130. Epub 2012 Oct 2. PMID 23037146
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419
- [Background] House WF, Hitselberger WE, Horn KL. The middle fossa transpetrous approach to the anterior-superior cerebellopontine angle. Am J Otol. 1986 Jan;7(1):1-4. PMID 3484905
- [Background] Mok J. HIV infection in children. J R Coll Gen Pract. 1988 Aug;38(313):342-4. No abstract available. PMID 3076903
- [Background] Pourtier-Piotte C, Pereira B, Soubrier M, Thomas E, Gerbaud L, Coudeyre E. French validation of the Foot Function Index (FFI). Ann Phys Rehabil Med. 2015 Oct;58(5):276-82. doi: 10.1016/j.rehab.2015.07.003. Epub 2015 Sep 4. PMID 26343763
- [Background] Kadri MA, Chevalier G, Mecheri H, Ngomo S, Lavalliere M, da Silva RA, Beaulieu LD. Time course and variability of tendinous vibration-induced postural reactions in forward and backward directions. J Electromyogr Kinesiol. 2020 Apr;51:102386. doi: 10.1016/j.jelekin.2020.102386. Epub 2020 Jan 20. PMID 32014802
- [Background] Hayashi K, Hirata Y, Kurushima H, Saeki M, Amioka H, Nomura S, Kuga Y, Ohkura Y, Ohtani H, Kajiyama G. Effect of dietary hydrogenated corn oil (trans-octadecenoate rich oil) on plasma and hepatic cholesterol metabolism in the hamster. Atherosclerosis. 1993 Feb;99(1):97-106. doi: 10.1016/0021-9150(93)90055-y. PMID 8461065